CLINICAL TRIAL: NCT05272930
Title: The Effect of Dionegest Use on the Frequency of Fibromyalgia in Endometriosis: A Cross-sectional Observational Study.
Brief Title: The Effect of Dionegest Use on the Frequency of Fibromyalgia in Endometriosis
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Fatma Ketenci Gencer, MD, Principal investigator, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpaşaTREHh
Record Dates: First submitted 2022-02-07; First posted 2022-03-10 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Fibromyalgia; Endometriosis Ovary; Dienogest
MeSH Terms: conditions — Fibromyalgia | interventions — dienogest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dienogest — Assessment of fibromyalgia effects after the use of dienogest

SUMMARY:
Endometriosis usually occurs during the reproductive period of women and poses a significant burden on quality of life and social costs. The estimated prevalence in premenopausal women is 10% in clinical studies and the frequency rises to 50% in symptomatic patients with pelvic pain and infertility. Observational studies in Europe estimated the prevalence to be 8-15 per 1000 people.

Fibromyalgia is a common musculoskeletal chronic painful condition that may be accompanied by cognitive impairment, somatic symptoms, fatigue, and psychiatric symptoms. The population frequency is given as 20-80 per 1000 people. Fibromyalgia is most often diagnosed in women aged 20-55 years; prevalence increases with age and is associated with a higher prevalence of comorbidities, including endocrine and genitourinary disorders. Co-existance of endometriosis and fibromyalgia is a special entity that has not been enlightened in detal yet.

DETAILED DESCRIPTION:
Although little is known about the causes of endometriosis, it is reported that women with endometriosis have a high rate of comorbidity with other chronic pain syndromes associated with peripheral and central changes in pain processing, including fibromyalgia, migraine headaches, inflammatory bowel disease, and painful bladder syndrome. Later, various studies conducted in different years showed that cross-organ sensitivity phenomenon, defined as the spread of harmful inputs (inflammation products, mediators, pathogens, etc.) from a diseased visceral organ to a normal organ, comorbidities including IBS, IBD, interstitial cystitis and chronic pelvic pain disorders are common. Therefore, it has been suggested that patients with endometriosis may have a higher risk of developing these chronic diseases. The results of another study are inconsistent with the studies that supports the coexistence of endometriosis and fibromyalgia.

These literature data indicate the need for more data on the frequency of fibromyalgia in women with endometriosis. On the other hand, it has been reported that pain scores are correlated with daily fluctuations of progesterone and testosterone in women with fibromyalgia, and progesterone and testosterone play a protective role for fibromyalgia pain. Dienogest is a fourth-generation selective progestin that has a significant local effect on endometriotic lesions, has little androgenic, less estrogenic, low glucocorticoid or mineralocorticoid activity and minimal effect on metabolic parameters, and is used in the medical treatment of endometriosis. However, there is no data on the effects of hormonal therapy used in the treatment of endometriosis on the frequency and severity of symptoms of fibromyalgia associated with endometriosis. Therefore, in this study, it was aimed to evaluate the effects of progesterone therapy used in endometriosis patients on fibromyalgia frequency, fibromyalgia severity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 40 years old
* Nulliparity
* Women diagnosed with endometrioma (unilateral, ≤ 4cm) by physical examination and vaginal/transabdominal ultrasonography

Exclusion Criteria:

* Pelvic mass that cannot be differentially diagnosed by physical examination and imaging techniques
* Endometrioma cases with surgical treatment indication
* Any concurrent major psychiatric disorder
* Any medical condition that may interfere with sensory perception (diabetes, neurological disorder, etc.)
* Presence of any other concomitant painful condition other than fibromyalgia and endometriosis
* Currently using any hormonal therapy
* History and/or presence of malignancy
* Pregnancy
* Menopause or premature ovarian failure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who applied to Gaziosmanpasa Training and Research Hospital Gynecology and Obstetrics Polyclinic, previously diagnosed with fibromyalgia and diagnosed with unilateral endometrioma.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Determination of recovery rate of participants diagnosed as in terms of fibromyalgia symptoms after dienogest use by using Visual Analog Scale (VAS). | 6 months
  VAS is a 10 cm labeled "No Pain" on one end and "The Most Severe Pain Possible" on the other. On a long line, the participant is asked to mark a point on this line that corresponds to the intensity of pain she feels. The distance between the starting point expressed as "No Pain" and the marked point is measured with a ruler and recorded in centimeters.
Determination of recovery rate of Symptom Severity (SS) Score in participants in terms of fibromyalgia symptoms after dienogest use by using Fibromyalgia Questionnaire Diagnostic Criteria and Symptom Severity Scale. | 6 months
  The first section contains 3 questions about fatigue, cognitive problems, and sleep symptoms, each scored in a likert format from 0 (no problem) to 3 (severe: persistent, life-disturbing problems) over the past week. The second part consists of 3 questions (maximum score 3) that give positive or negative answers to the following somatic complaints that have arisen in the last 6 months; abdominal pain or cramps, depression and headache. The sum of Parts 1 and 2 provides a Symptom Severity (SS) Score in the range of 0-12.
Determination of recovery rate of Widespread Pain Index (WPI) Score in participants in terms of fibromyalgia symptoms after dienogest use by using Fibromyalgia Questionnaire Diagnostic Criteria and Symptom Severity Scale | 6 months
  The third section is a measurement of the Widespread Pain Index (WPI) and is completed by identifying body areas where pain or tenderness has been felt during the previous 7 days. The maximum score for the WPI section is 19. Polysymptomatic distress (PSD) is defined as the sum of the (0-19) WPI and the 6-item (0-12) SS scale, ranging from 0-31.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No